CLINICAL TRIAL: NCT03072134
Title: Neural Stem Cell Oncolytic Adenoviral Virotherapy of Newly Diagnosed Malignant Glioma
Brief Title: Neural Stem Cell Based Virotherapy of Newly Diagnosed Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Maciej Lesniak, Professor and Chairman, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00203933; 5P50CA221747-05 (NIH)
Record Dates: First submitted 2017-02-20; First posted 2017-03-07 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Glioma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma; Glioblastoma Multiforme; Astrocytoma, Grade III; Astrocytoma, Grade IV; Brain Cancer
Keywords: Glioma; Glioblastoma; Astrocytoma; Brain Cancer; New Diagnosed Glioma; Temozolomide; Radiation; Neural Stem Cells; Virotherapy; Adenovirus; Oncolytic virotherapy
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma; Brain Neoplasms; Adenoviridae Infections

STUDY DESIGN:
Intervention Model Description: A Phase I study of neural stem cell based virotherapy in combination with standard radiation and chemotherapy for patients with newly diagnosed malignant glioma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Unresectable disease (Experimental): Patients with unresectable tumors will undergo a biopsy followed by injection of neural stem cells loaded with the virus and then receive standard chemoradiotherapy.
  Interventions: Biological: Neural stem cells loaded with an oncolytic adenovirus
- Resectable disease (Experimental): Patients with resectable tumors will undergo a resection followed by injection of neural stem cells loaded with the virus and then receive standard chemoradiotherapy.
  Interventions: Biological: Neural stem cells loaded with an oncolytic adenovirus

INTERVENTIONS:
Biological: Neural stem cells loaded with an oncolytic adenovirus — The primary objectives are to evaluate the safety of the combined therapy and determine the maximum tolerated dose (MTD) for a future Phase II study.
  Other Names: NSC-CRAd-Survivin-pk7

SUMMARY:
Malignant gliomas have a very poor prognosis with median survival measured in months rather than years. It is a disease in great need of novel therapeutic approaches. Based on the encouraging results of our preclinical studies which demonstrate improved efficacy without added toxicity, the paradigm of delivering a novel oncolytic adenovirus via a neural stem cell line in combination with radiation and chemotherapy is well-suited for evaluation in newly diagnosed malignant gliomas. The standard-of-care allows application of virotherapy as neoadjuvant therapy and assessment of the cooperative effects with radiation/chemotherapy without altering the standard treatment.

DETAILED DESCRIPTION:
This is an open-label, phase 1, dose escalation trial that followed a 3x3 design. Three doses will be evaluated in the resectable cohorts: Cohort 1: 0.5x10^8 NSCs loading 6.25x10^10 vp; Cohort 2: 1.0x10^8 NSCs loading 1.25x10^11 vp; and Cohort 3: 1.5x10^8 NSCs loading 1.875x10^11 vp. Subjects enrolled have newly diagnosed high-grade glioma based on clinical and radiologic criteria; pathology will be confirmed at the time of surgical resection. Direct intra-tumoral injection of study product (NSC-CRAd-S-p7) will be done after resection but prior to closure. Subjects will then receive concomitant radiotherapy (RT) at a dose of 60Gy and chemotherapy with temozolomide (TMZ), 75 mg/m2, daily during RT. This will be followed by adjuvant TMZ dosed at 200 mg/m2 for 6 cycles. Subjects will be followed until disease progression with serial brain MRIs, and for survival up to 5 years. The non-resectable cohort will not opened due to limited product availability.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have presumed malignant glioma based on clinical and radiologic evaluation (pathologic confirmation of malignant glioma must be made at the time of stereotactic biopsy or resection prior to NSC-CRAd-S-pk7 injection; if this is not possible, the injection will not be performed and the subject will no longer be eligible for the study).
* Tumor must be accessible for injection and must not be located in the brainstem, or contained within the ventricular system.
* Planning to undergo standard radiation/chemotherapy
* 18 years of age or older.
* Performance status must be KPS ≥ 70
* SGOT (AST) < 3x upper limit of normal
* Serum creatinine < 2mg/dl
* Platelets > 100,000/mm3 and WBC > 3000/mm3

Exclusion Criteria:

* Prior or ongoing liver disease including known cirrhosis, hepatitis B or C infection but not to exclude patients with a distant history of resolved hepatitis A infection.
* Immunosuppressive drugs (with exception of corticosteroid).
* Known HIV+ patients.
* Acute infections (viral, bacterial or fungal infections requiring therapy).
* Pregnant or breast-feeding patients.
* Evidence of metastatic disease or other malignancy (except squamous or basal cell skin cancers).
* Prior radiation therapy to the brain or prior treatment for brain tumor Other serious co-morbid illness or compromised organ function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej S Lesniak, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Northwestern Memorial Hospital, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tobias AL, Thaci B, Auffinger B, Rincon E, Balyasnikova IV, Kim CK, Han Y, Zhang L, Aboody KS, Ahmed AU, Lesniak MS. The timing of neural stem cell-based virotherapy is critical for optimal therapeutic efficacy when applied with radiation and chemotherapy for the treatment of glioblastoma. Stem Cells Transl Med. 2013 Sep;2(9):655-66. doi: 10.5966/sctm.2013-0039. Epub 2013 Aug 7. PMID 23926209
- [Background] Ahmed AU, Thaci B, Tobias AL, Auffinger B, Zhang L, Cheng Y, Kim CK, Yunis C, Han Y, Alexiades NG, Fan X, Aboody KS, Lesniak MS. A preclinical evaluation of neural stem cell-based cell carrier for targeted antiglioma oncolytic virotherapy. J Natl Cancer Inst. 2013 Jul 3;105(13):968-77. doi: 10.1093/jnci/djt141. PMID 23821758
- [Background] Ahmed AU, Tyler MA, Thaci B, Alexiades NG, Han Y, Ulasov IV, Lesniak MS. A comparative study of neural and mesenchymal stem cell-based carriers for oncolytic adenovirus in a model of malignant glioma. Mol Pharm. 2011 Oct 3;8(5):1559-72. doi: 10.1021/mp200161f. Epub 2011 Jun 30. PMID 21718006
- [Background] Ahmed AU, Thaci B, Alexiades NG, Han Y, Qian S, Liu F, Balyasnikova IV, Ulasov IY, Aboody KS, Lesniak MS. Neural stem cell-based cell carriers enhance therapeutic efficacy of an oncolytic adenovirus in an orthotopic mouse model of human glioblastoma. Mol Ther. 2011 Sep;19(9):1714-26. doi: 10.1038/mt.2011.100. Epub 2011 May 31. PMID 21629227
- [Background] Ulasov IV, Sonabend AM, Nandi S, Khramtsov A, Han Y, Lesniak MS. Combination of adenoviral virotherapy and temozolomide chemotherapy eradicates malignant glioma through autophagic and apoptotic cell death in vivo. Br J Cancer. 2009 Apr 7;100(7):1154-64. doi: 10.1038/sj.bjc.6604969. Epub 2009 Mar 10. PMID 19277041
- [Background] Nandi S, Ulasov IV, Tyler MA, Sugihara AQ, Molinero L, Han Y, Zhu ZB, Lesniak MS. Low-dose radiation enhances survivin-mediated virotherapy against malignant glioma stem cells. Cancer Res. 2008 Jul 15;68(14):5778-84. doi: 10.1158/0008-5472.CAN-07-6441. PMID 18632631
- [Background] Ulasov IV, Zhu ZB, Tyler MA, Han Y, Rivera AA, Khramtsov A, Curiel DT, Lesniak MS. Survivin-driven and fiber-modified oncolytic adenovirus exhibits potent antitumor activity in established intracranial glioma. Hum Gene Ther. 2007 Jul;18(7):589-602. doi: 10.1089/hum.2007.002. PMID 17630837
- [Derived] Fares J, Ahmed AU, Ulasov IV, Sonabend AM, Miska J, Lee-Chang C, Balyasnikova IV, Chandler JP, Portnow J, Tate MC, Kumthekar P, Lukas RV, Grimm SA, Adams AK, Hebert CD, Strong TV, Amidei C, Arrieta VA, Zannikou M, Horbinski C, Zhang H, Burdett KB, Curiel DT, Sachdev S, Aboody KS, Stupp R, Lesniak MS. Neural stem cell delivery of an oncolytic adenovirus in newly diagnosed malignant glioma: a first-in-human, phase 1, dose-escalation trial. Lancet Oncol. 2021 Aug;22(8):1103-1114. doi: 10.1016/S1470-2045(21)00245-X. Epub 2021 Jun 29. PMID 34214495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 24, 2017 thru Nov 13, 2019 at Northwestern University and City of Hope.
Pre-assignment Details: Arm A, for subjects with unresectable disease, was not opened due to limited product availability
Groups:
- Resectable Disease: Patients with resectable tumors will undergo a resection followed by injection of neural stem cells loaded with the virus and then receive standard chemoradiotherapy. The unresectable cohort was not able to be opened due to limited product availability.
  Neural stem cells loaded with an oncolytic adenovirus: The primary objectives are to evaluate the safety of the combined therapy and determine the maximum tolerated dose (MTD) for a future Phase II study.
Period: Cohort 1: 0.5x10^8/NSCs/6.25x10^10 vp
Arm/Group | Resectable Disease
Started | 3
Completed | 3
Not Completed | 0
Period: Cohort 2: 1.0x10^8 NSCs/1.25x10^10 vp
Arm/Group | Resectable Disease
Started | 3
Completed | 3
Not Completed | 0
Period: Cohort 3: 1.5x10^8 NSCs/1.875x10^10 vp
Arm/Group | Resectable Disease
Started (An additional 3 subjects were added as one subject at this dose level experienced a DLT.) | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B: Resectable Disease Cohort 1: Patients with resectable tumors will undergo a resection followed by injection of neural stem cells loaded with the virus at dose level 0.5x10^8 NSCs loading 6.25x10^10 vp and then receive standard chemoradiotherapy.
  Neural stem cells loaded with an oncolytic adenovirus: The primary objectives are to evaluate the safety of the combined therapy and determine the maximum tolerated dose (MTD) for a future Phase II study.
- Arm B: Resectable Disease Cohort 2: Patients with resectable tumors will undergo a resection followed by injection of neural stem cells loaded with the virus at dose level 1.0x10^8 NSCs loading 1.25x10^11 vp and then receive standard chemoradiotherapy.
  Neural stem cells loaded with an oncolytic adenovirus: The primary objectives are to evaluate the safety of the combined therapy and determine the maximum tolerated dose (MTD) for a future Phase II study.
- Arm B: Resectable Disease Cohort 3: Patients with resectable tumors will undergo a resection followed by injection of neural stem cells loaded with the virus at dose level 1.5x10^8 NSCs loading 1.875x10^11 vp and then receive standard chemoradiotherapy.
  Neural stem cells loaded with an oncolytic adenovirus: The primary objectives are to evaluate the safety of the combined therapy and determine the maximum tolerated dose (MTD) for a future Phase II study.
- Total: Total of all reporting groups
Arm/Group | Arm B: Resectable Disease Cohort 1 | Arm B: Resectable Disease Cohort 2 | Arm B: Resectable Disease Cohort 3 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants] — Adult Population
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 3 | 3 | 6 | 12
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 1 | 1 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 3 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Dose-limiting Toxicities
Description: Using a 3+3 dose escalation design, three to six patients were to be enrolled per dose in each of the 3 cohorts. If no patients in the cohort experienced a dose-limiting toxicity (DLT), then the next cohort enrolled a minimum of 3 patients. If one of three patients experienced a DLT, then 3 more patients were evaluated at that dose level. If none of these three additional patients experienced a DLT, then dose escalation occurs, unless this is the highest dose, in which case dose escalation is stopped and the highest dose is declared the MTD. If 1 or more of these additional 3 patients had a DLT, then three additional patients may be entered, after discussion with the sponsor, at the next lowest does level if only three patients were treated previously at that dose. If two or more patients experienced a DLT Dose escalation will be stopped; 3 more patients could be added with sponsor approval at the next lower dose level.
Time Frame: Two years
Population: No screen failures were encountered and all 12 patients were evaluable.
Measure: Number; unit: Percentage of dose-limiting toxicities
Groups:
- Arm B/Cohort 1: Patients with resectable tumors will undergo a resection followed by injection of neural stem cells loaded with the virus (dose: 0.5x10^8/NSCs/6.25x10^10 vp) and then receive standard chemoradiotherapy. No dose limiting toxicities were experienced in this cohort.
- Arm B/Cohort 2: Patients with resectable tumors will undergo a resection followed by injection of neural stem cells loaded with the virus (dose: 1.0x10^8 NSCs/1.25x10^10 vp) and then receive standard chemoradiotherapy. No dose limiting toxicities were experienced in this cohort.
- ArmB/Cohort 3: .5x10^8 NSCs/1.875x10^10 vp
  Patients with resectable tumors will undergo a resection followed by injection of neural stem cells loaded with the virus (dose: 1.5x10^8 NSCs/1.875x10^10 vp) and then receive standard chemoradiotherapy. One dose limiting toxicity event was experienced in this cohort, prompting 3 additional patients being added to the cohort; no dose limiting toxicities were experienced in this addition to the cohort, and this dose was determined to be the MTD.
Arm/Group | Arm B/Cohort 1 | Arm B/Cohort 2 | ArmB/Cohort 3
Number analyzed (Participants) | 3 | 3 | 6
Percentage of dose-limiting toxicities | 0 | 0 | 17

2. Secondary Outcome: Assessment of Tumor Response.
Description: Per Response Assessment in Neuro-Oncology Criteria (RANO, 2017) for target lesions as assessed by MRI: Complete Response (CR): The enhancing tumor is no longer seen by neuroimaging; Partial Response (PR): Decrease of ≥ 50% in the product of two diameters with the patient on a stable or decreasing dose of steroids; Minor Response (MR): Decrease in diameter products of < 50% with the patient on a stable or decreasing dose of steroids; Stable Disease (SD): The scan shows no change. Patients should be receiving stable or decreasing doses of steroids; Progression (P): Increase of > 25% in tumor area (two diameters) provided that the patient has not had his/her dose of steroids decreased since the last evaluation period. A concomitant decrease in steroid dose will rule out a progression designation during the first two months after completion of radiation; Pseudoprogression (PP): Radiological changes without concomitant neurological changes.
Time Frame: Two years
Population: Nine of 12 patients had measureable disease post-surgery and were followed with serial MRIs.
Measure: Number; unit: Percentage of participants
Groups:
- Total Cohort: Analyses were conducted for the entire cohort (N=12) for secondary objectives.
Arm/Group | Total Cohort
Number analyzed (Participants) | 12
Percentage of participants
  Percentage of participants with tumor response: Partial | 8
  Percentage of participants with tumor response: Pseudoprogression | 8
  Percentage of participants with tumor response: Stable disease | 84

3. Secondary Outcome: Progression-free Survival
Description: Median progression-free survival
Time Frame: two years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total Cohort
Number analyzed (Participants) | 12
Months | 9.1 [8.5 to 36]

4. Secondary Outcome: Overall Survival
Description: Median overall survival
Time Frame: Two years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total Cohort
Number analyzed (Participants) | 12
Months | 18.4 [6.5 to 36]

ADVERSE EVENTS:
Time Frame: Two years and 7 months
Description: Number of patients in each cohort affected by serious adverse events
Groups:
- Resectable Disease Cohort 1: Patients with resectable tumors underwent surgical resection followed by injection of neural stem cells loaded with the virus (0.5x10^8 NSCs loading 6.25x10^10 vp) and then received standard chemoradiotherapy.
- Resectable Disease Cohort 2: Patients with resectable tumors underwent surgical resection followed by injection of neural stem cells loaded with the virus (.0x10^8 NSCs loading 1.25x10^11 vp) and then received standard chemoradiotherapy.
- Resectable Disease Cohort 3: Patients with resectable tumors underwent surgical resection followed by injection of neural stem cells loaded with the virus (1.5x10^8 NSCs loading 1.875x10^11 vp) and then received standard chemoradiotherapy.
Arm/Group | Resectable Disease Cohort 1 | Resectable Disease Cohort 2 | Resectable Disease Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resectable Disease Cohort 1 (N=3) | Resectable Disease Cohort 2 (N=3) | Resectable Disease Cohort 3 (N=6)
Meningitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Viral meningitis
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Edema, cerebral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resectable Disease Cohort 1 (N=3) | Resectable Disease Cohort 2 (N=3) | Resectable Disease Cohort 3 (N=6)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 3 (7)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (3)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2)
Fatigue (General disorders) | 3 (4) | 1 (2) | 2 (4)
Malaise (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (7) | 3 (8) | 5 (8)
Platelet count decreased (Investigations) | 2 (3) | 1 (1) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 3 (5) | 6 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5) | 2 (2) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 2 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (5) | 6 (10)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 3 (3)
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 3 (6) | 5 (11)
Thromboembolic event (Vascular disorders) | 2 (4) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (2) | 1 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dermatitis, radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders, other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Subdural fluid collection
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03072134/Prot_SAP_000.pdf